CLINICAL TRIAL: NCT00681486
Title: Ghrelin - A Possible Opportunity to Improve Appetite, Nutritional State, Metabolic Integrity and Physical Functioning in Cancer Patients With Progressive Weight Loss
Brief Title: Ghrelin - A Possible Opportunity to Improve Appetite
Acronym: Phase 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Swedish Cancer Foundation (Other); Medical Research Council (Other Government)
Responsible Party: Professor Kent Lundholm, University of Gothenburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: kl4501123
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Cancer
Keywords: Ghrelin; Nutrition; Cancer patients; Survival
MeSH Terms: conditions — Neoplasms | interventions — Ghrelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- A, 1 (Active Comparator): Ghrelin
  Interventions: Drug: Ghrelin
- A, 2 (Active Comparator): Ghrelin.
  Interventions: Drug: Ghrelin

INTERVENTIONS:
Drug: Ghrelin — High dose of ghrelin given as subcutaneous injection once a day for the duration of 8 weeks.
  Arms: A, 1
Drug: Ghrelin — Low dose of ghrelin given as subcutaneous injection once a day for the duration of 8 weeks.
  Arms: A, 2

SUMMARY:
The study is designed to evaluate whether ghrelin treatment can improve appetite in weight losing cancer patients.

DETAILED DESCRIPTION:
Randomized study with follow up evaluations each month until preterminal state. Cancer patients will be randomised to either high dose or low dose of active treatment given as daily injection.

ELIGIBILITY:
Inclusion Criteria:

* Weight loss

Exclusion Criteria:

* Diabetes

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-10; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Food intake | June 2008

CONTACTS AND LOCATIONS:
Overall Officials: Kent Lundholm, MD, prof, Principal Investigator — Göteborg University
Locations (1):
- Department of surgery, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- See also: Göteborg University — http://gu.se